CLINICAL TRIAL: NCT04375891
Title: Randomized Phase II Study of Radiation Therapy Alone Versus Radiation Therapy Plus Radiofrequency Ablation (RFA)/Vertebral Augmentation for Localized Spine Metastasis
Brief Title: Radiation Therapy Alone Versus Radiation Therapy Plus Radiofrequency Ablation (RFA)/Vertebral Augmentation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-KOT-001
Record Dates: First submitted 2020-03-13; First posted 2020-05-06 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Oncology; Spine Metastases
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy; Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: A study design of 2:1 randomization scheme (RT plus PVA/RFA:RT), the study will be adequately powered with 52 patients (35 in the RT plus PVA/RFA arm and 17 in the RT arm). Assuming a 5% ineligibility rate, a death rate of 15%, and a patient non-compliance rate of 15%, the total sample size required would be 80 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy (Other): Radiotherapy alone
  Interventions: Radiation: Radiation Therapy
- Radiotherapy plus radiofrequency ablation (Other): Radiotherapy plus radiofrequency ablation / vertebral augmentation(Combination therapy)
  Interventions: Radiation: Radiation Therapy; Radiation: Radiofrequency Ablation (RFA)

INTERVENTIONS:
Radiation: Radiation Therapy — 30 Gy in 10 fractions of 3 Gy each
Radiation: Radiofrequency Ablation (RFA) — Radiofrequency Ablation (RFA) / Vertebral Augmentation
  Arms: Radiotherapy plus radiofrequency ablation

SUMMARY:
The spread of cancer to the spine is referred to as spine metastasis. Spine metastases are a common complication of cancer and are frequently associated with significant back pain. This study is being done to help improve treatment for back pain caused by spinal metastases by comparing the effectiveness of two standard treatments. These two treatments include radiation therapy (RT) alone versus radiation therapy combined with radiofrequency ablation, with or without vertebral augmentation (PVA/RFA). In addition to RT or RT with PVA/RFA, will be continued with current pain medications.

DETAILED DESCRIPTION:
All supportive therapy for optimal medical care will be given during the study period at the discretion of the attending physician(s) within the parameters of the protocol and documented on each site's source documents as concomitant medication.

The study will be adequately powered with 52 patients (35 in the RT plus PVA/RFA arm and 17 in the RT arm). Assuming a 5% ineligibility rate, a death rate of 15%, and a patient non-compliance rate of 15%, the total sample size required would be 80 patients.

Patients will be stratified according to the tumor type (radioresistant [soft tissue sarcoma, melanoma, and renal cell carcinoma] versus other types). The treatment allocation scheme described by Zelen (1974) will be used because it balances patient factors. Within each stratum, patients will be randomized in a 2:1 ratio to either image-guided RT plus RFA/PVA or external beam RT alone.

The 2:1 randomization allocation will be used to accommodate increased demand for image-guided RT plus RFA/PVA.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have localized spine metastasis from the T5 to L5 levels by an imaging study (bone scan, PET, CT, or MRI). Patients can have other visceral metastasis, and radioresistant tumors (including soft tissue sarcomas, melanomas, and renal cell carcinomas) are eligible.
* Zubrod Performance Status 0-3
* History/physical examination within 2 weeks prior to registration
* Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential; Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control;
* MRI (contrast is not required but strongly recommended) of the involved spine within 6 weeks prior to registration to determine the extent of the spine involvement;
* Numerical Rating Pain Scale within 1 week prior to registration; the patient must have a score on the Scale of ≥ 5 for at least one of the planned sites for intervention. Documentation of the patient's initial pain score is required. Patients taking medication for pain at the time of registration are eligible.
* Patients with epidural compression are eligible provided that there is a ≥ 3 mm gap between the spinal cord and the edge of the epidural lesion.
* Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

* Histologies of myeloma, lymphoma, small-cell lung cancer, germ-cell tumor
* Non-ambulatory patients;
* Frank spinal cord compression or displacement or epidural compression within 3 mm of the spinal cord;
* Patients with rapid neurologic decline;
* Bony retropulsion causing neurologic abnormality;
* Prior radiation to the index spine
* Patients requiring immediate neurosurgical intervention
* Patients receiving concurrent chemotherapy
* Patients needing palliative to more than 2 sites of spinal disease in total

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in pain control | 3 months, 6, 12, 24 months
  Change in pain control (as measured by the 11 point Numeric pain rating scale) as compared to conventional palliative radiotherapy alone.

SECONDARY OUTCOMES:
Change in pain response | 3 months, 6, 12, 24 months
  Change in the rapidity of pain response at the treated site(s) as compared to conventional Radiotherapy alone, as measured by the Numeric pain rating scale.
Measure increases in the duration of pain response | 3 months, 6, 12, 24 months
  Measure increases in the duration of pain response at the treated site(s), as compared to conventional RT alone, as measured by the Numeric pain rating scale.
Number of adverse events | 3 months, 6, 12, 24 months
  Number of adverse events between the two treatments according to the NCI Common Terminology Criteria for Adverse Events version 5.0.
Measure the potential benefit on quality of life | 3 months, 6, 12, 24 months
  Measure the potential benefit of radiotherapy plus Vertebral Augmentation/Radiofrequency Ablation on change in and overall quality of life, as measured by the Functional Assessment of Cancer Therapy-General; in pain as measured by the Brief Pain Inventory; and in health utilities as measured by the EuroQol

CONTACTS AND LOCATIONS:
Overall Officials: Rupesh Kotecha, MD, Principal Investigator — Miami Cancer Institute (MCI) at Baptist Health South Florida
Locations (1):
- Miami Cancer Institute at Baptist Health South Florida, Miami, Florida, United States

REFERENCES:
- [Derived] Kotecha R, Schiro BJ, Sporrer J, Rubens M, Appel HR, Calienes KS, Boulanger B, Pujol MV, Suarez DT, Pena A, Kudryashev A, Mehta MP. Radiation therapy alone versus radiation therapy plus radiofrequency ablation/vertebral augmentation for spine metastasis: study protocol for a randomized controlled trial. Trials. 2020 Nov 23;21(1):964. doi: 10.1186/s13063-020-04895-x. PMID 33228756
- See also: Miami Cancer Institute website — http://baptisthealth.net/cancer-care/home